CLINICAL TRIAL: NCT01347216
Title: Prospective Registry of Newly Initiated Therapies for Pulmonary Hypertension
Brief Title: COMPERA / COMPERA-KIDS
Acronym: COMPERA
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: COMPERA
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Hypertension (PH)
Keywords: Drug treatment; Treatment pathways; Clinical routine; Registry; Treatment outcomes; Endothelin receptor antagonist; Phosphodiesterase-V inhibitor; Prostanoid; Sildenafil; Bosentan; Macitentan; Sitaxentan; Ambrisentan; Imatinib; Epoprostenol; Treprostinil; Iloprost; Infusion pump; Riociguat; soluble guanylate cyclase stimulator; Quality of life; Patient-related outcomes; Economic model; Adverse event; Safety; Combination therapy; Internet; Europe; Eisenmenger; Adults; Children; Selexipag; Baltic states; Risk
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Eisenmenger Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In view of the manifold options for mono- and combination therapy that have now emerged for patients with pulmonary (arterial) hypertension (PH/PAH), controlled clinical trials can only provide part of the information needed for optimal management. In order to gather adequate data on PAH/PH treatment in routine clinical care, the ongoing COMPERA registry prospectively documents consecutive patients with newly initiated treatment of PAH/PAH since May 2007. The internet-based registry fulfills high quality standards through several measures (planned minimum centre contribution of at least 10 patients per year, automated plausibility checks of data at entry, queries, monitoring with source data verification in >50% of participating centers). It can be applied, among further purposes, for quality assurance: individual centers can confidentially compare their results with the combined outcome of other centers and the recommendations from guidelines. It is expected that the register contributes to optimization of specific drug therapy for PAH and PH.

Since July 2013, also children of any age can be documented (COMPERA-KIDS).

DETAILED DESCRIPTION:
COMPERA will report current and comprehensive data on

* Demographics and clinical course of incident and prevalent PAH and PH patients
* Patient outcomes including survival, by subgroup, by treatment strategy and other factors
* Clinical predictors of short-term and long-term clinical outcomes
* Relationship between PAH medications and patient outcomes
* Temporal trends in treatments and outcomes for newly diagnosed patients
* The state of implementation of current PAH guidelines
* Evolving research needs of the PAH community
* Patients with PAH associated with congenital heart disease and Eisenmenger physiology who do not receive specific drug therapy for PAH ("COMPERA-Eisenmenger", as stated in the amendment dated 23. January 2012).
* Children of any age with PH or PAH (all Dana Point groups), as stated in the amendment dated 1 June 2013 ("COMPERA-KIDS").

ELIGIBILITY:
Inclusion Criteria:

* All age groups (amendment dated 1 June 2013)
* Written informed consent
* Pulmonary hypertension (PH) of either

  * PAH: idiopathic form (IPAH) or
  * PAH associated with connective tissue diseases (PAH-CTD), with congenital heart defects (PAH-CHD), with HIV infection (PAH-HIV), or the portopulmonary form
  * Chronic thromboembolic PH (CTEPH)
  * PH in left heart diseases (with isolated diastolic dysfunction; with systolic dysfunction, other)
  * PH in pulmonary disease (chronic obstructive pulmonary disease; interstitial fibrosis, etc.)
  * "Relative PH" in CHD after cavopulmonary anastomosis or Fontan-type surgery, even without the classical pulmonary pressure criteria of PH.
* Newly initiated (i.e. a maximum of 3 months before documentation for the first time) therapy with endothelin receptor antagonists (ERA), phoshodiesterase-5 (PDE-5) inhibitors, soluble guanylate cyclase (sGC) stimulators or prostacyclins in mono- or combination therapy.

Exceptions: PAH-CHD patients can be included on maintenance or newly initiated PAH therapy (3-month rule dose not apply).

PAH-CHD patients with severe pulmonary vascular disease (e.g. Eisenmenger physiology) irrespective of treatment with any PAH drugs are eligible for inclusion, too.

Exclusion Criteria:

* Patients on maintenance therapy, i.e. previous treatment with any ERA/ PDE-5 inhibitor/prostacyclin/sGC stimulator drug longer than 3 months before documentation for the first time (exception: PAH-CHD patients).

Min Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any manifestation of pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2007-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients on monotherapy vs combination therapies at baseline and during follow-up (drug utilisation patterns) | Up to 10 years after inclusion

SECONDARY OUTCOMES:
Number of patients in the various Dana Point groups (patient characteristics in PAH and non-PAH pulmonary hypertension groups) | Up to 10 years after inclusion
Probability of survival in the various Dana Point groups (PAH and non-PAH pulmonary hypertension groups) by Kaplan-Meier estimate | Up to 10 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marius M Hoeper, MD, PhD, Principal Investigator — Department of Pulmonology, Medical School Hannover, Germany; Ardeschir H. Ghofrani, MD, PhD, Study Director — Lung Centre, Giessen, Germany; Marion Delcroix, MD, PhD, Study Director — Dept of Pneumology, University Leuven, Belgium; Dario Vizza, MD, PhD, Study Director — Department of Cardiovascular and Respiratory Sciences, University La Sapienza, Rome, Italy; David Pittrow, MD, PhD, Study Director — Institute for Clinical Pharmacoloy, Medical Faculty, Technical University Dresden, Germany; Christian Opitz, MD, PhD, Study Director — Department of Cardiology, DRK-Kliniken Berlin, Germany; Oliver Distler, MD, PhD, Study Director — Department for Rheumatology, University Hospital Zurich, Switzerland; Harald Kaemmerer, MD, PhD, Study Director — German Heart Centre, Munich, Germany; Stephan Rosenkranz, MD, PhD, Study Director — Heart Centre, Cologne; Ekkehard Grünig, MD, PhD, Study Director — Centre for Pulmonary Hypertension at Thoraxclinic Heidelberg, Germany; Matthias Gorenflo, MD, PhD, Principal Investigator — Dept. Paed. Cardiol./Congenital Cardiology, Heidelberg University Medical Centre, Germany; Karen Olsson, MD, PhD, Study Director — Department of Pulmonology, Medical School Hannove
Locations (7):
- Dept. of Pneumology, University, Leuven, Belgium
- Germany (4):
  - DRK-Klinikum Köpenick, Berlin
  - Lung Centre, University of Giessen, Giessen
  - Department of Pulmology; Hannover Medical School, Hanover
  - German Heart Centre, Munich
- Department of Cardiovascular and Respiratory Sciences, University La Sapienza, Rome, Italy
- Dept. for Rheumatology, University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data sharing has not been planned.

REFERENCES:
- [Background] Pausch C, Pittrow D, Hoeper MM, Huscher D. Performance of the ESC/ERS 4-strata risk stratification model for pulmonary arterial hypertension with missing variables. Eur Respir J. 2023 Nov 29;62(5):2301023. doi: 10.1183/13993003.01023-2023. Print 2023 Nov. PMID 37802633
- [Background] Pittrow D, Ghofrani HA, Opitz CF, Huscher D, Hoeper MM. [International, prospective register for the documentation of first-line and maintenance therapy in patients with pulmonary hypertension (CompERA-XL)]. Dtsch Med Wochenschr. 2009 Aug;134 Suppl 5:S173-5. doi: 10.1055/s-0029-1225318. Epub 2009 Aug 28. German. PMID 19718609
- [Background] Hoeper MM, Huscher D, Ghofrani HA, Delcroix M, Distler O, Schweiger C, Grunig E, Staehler G, Rosenkranz S, Halank M, Held M, Grohe C, Lange TJ, Behr J, Klose H, Wilkens H, Filusch A, Germann M, Ewert R, Seyfarth HJ, Olsson KM, Opitz CF, Gaine SP, Vizza CD, Vonk-Noordegraaf A, Kaemmerer H, Gibbs JS, Pittrow D. Elderly patients diagnosed with idiopathic pulmonary arterial hypertension: results from the COMPERA registry. Int J Cardiol. 2013 Sep 30;168(2):871-80. doi: 10.1016/j.ijcard.2012.10.026. Epub 2012 Nov 17. PMID 23164592
- [Background] Olsson KM, Delcroix M, Ghofrani HA, Tiede H, Huscher D, Speich R, Grunig E, Staehler G, Rosenkranz S, Halank M, Held M, Lange TJ, Behr J, Klose H, Claussen M, Ewert R, Opitz CF, Vizza CD, Scelsi L, Vonk-Noordegraaf A, Kaemmerer H, Gibbs JS, Coghlan G, Pepke-Zaba J, Schulz U, Gorenflo M, Pittrow D, Hoeper MM. Anticoagulation and survival in pulmonary arterial hypertension: results from the Comparative, Prospective Registry of Newly Initiated Therapies for Pulmonary Hypertension (COMPERA). Circulation. 2014 Jan 7;129(1):57-65. doi: 10.1161/CIRCULATIONAHA.113.004526. Epub 2013 Sep 30. PMID 24081973
- [Background] Kramm T, Wilkens H, Fuge J, Schafers HJ, Guth S, Wiedenroth CB, Weingard B, Huscher D, Pittrow D, Cebotari S, Hoeper MM, Mayer E, Olsson KM. Incidence and characteristics of chronic thromboembolic pulmonary hypertension in Germany. Clin Res Cardiol. 2018 Jul;107(7):548-553. doi: 10.1007/s00392-018-1215-5. Epub 2018 Feb 15. PMID 29450722
- [Background] Hoeper MM, Kramer T, Pan Z, Eichstaedt CA, Spiesshoefer J, Benjamin N, Olsson KM, Meyer K, Vizza CD, Vonk-Noordegraaf A, Distler O, Opitz C, Gibbs JSR, Delcroix M, Ghofrani HA, Huscher D, Pittrow D, Rosenkranz S, Grunig E. Mortality in pulmonary arterial hypertension: prediction by the 2015 European pulmonary hypertension guidelines risk stratification model. Eur Respir J. 2017 Aug 3;50(2):1700740. doi: 10.1183/13993003.00740-2017. Print 2017 Aug. PMID 28775047
- [Background] Hoeper MM, Pittrow D, Opitz C, Gibbs JSR, Rosenkranz S, Grunig E, Olsson KM, Huscher D. Risk assessment in pulmonary arterial hypertension. Eur Respir J. 2018 Mar 29;51(3):1702606. doi: 10.1183/13993003.02606-2017. Print 2018 Mar. No abstract available. PMID 29599117
- [Background] Zelniker TA, Huscher D, Vonk-Noordegraaf A, Ewert R, Lange TJ, Klose H, Dumitrescu D, Halank M, Held M, Gall H, Pittrow D, Hoeper MM, Frankenstein L. The 6MWT as a prognostic tool in pulmonary arterial hypertension: results from the COMPERA registry. Clin Res Cardiol. 2018 Jun;107(6):460-470. doi: 10.1007/s00392-018-1207-5. Epub 2018 Jan 24. PMID 29368137
- [Background] Delcroix M, Staehler G, Gall H, Grunig E, Held M, Halank M, Klose H, Vonk-Noordegraaf A, Rosenkranz S, Pepke-Zaba J, Opitz CF, Gibbs JSR, Lange TJ, Tsangaris I, Huscher D, Pittrow D, Olsson KM, Hoeper MM. Risk assessment in medically treated chronic thromboembolic pulmonary hypertension patients. Eur Respir J. 2018 Nov 8;52(5):1800248. doi: 10.1183/13993003.00248-2018. Print 2018 Nov. PMID 30337446
- [Background] Kaemmerer H, Gorenflo M, Huscher D, Pittrow D, Apitz C, Baumgartner H, Berger F, Bruch L, Brunnemer E, Budts W, Claussen M, Coghlan G, Dahnert I, D'Alto M, Delcroix M, Distler O, Dittrich S, Dumitrescu D, Ewert R, Faehling M, Germund I, Ghofrani HA, Grohe C, Grossekreymborg K, Halank M, Hansmann G, Harzheim D, Nemes A, Havasi K, Held M, Hoeper MM, Hofbeck M, Hohenfrost-Schmidt W, Jureviciene E, Gumbiene L, Kabitz HJ, Klose H, Kohler T, Konstantinides S, Koestenberger M, Kozlik-Feldmann R, Kramer HH, Kropf-Sanchen C, Lammers A, Lange T, Meyn P, Miera O, Milger-Kneidinger K, Neidenbach R, Neurohr C, Opitz C, Perings C, Remppis BA, Riemekasten G, Scelsi L, Scholtz W, Simkova I, Skowasch D, Skride A, Stahler G, Stiller B, Tsangaris I, Vizza CD, Vonk Noordegraaf A, Wilkens H, Wirtz H, Diller GP, Grunig E, Rosenkranz S. Pulmonary Hypertension in Adults with Congenital Heart Disease: Real-World Data from the International COMPERA-CHD Registry. J Clin Med. 2020 May 13;9(5):1456. doi: 10.3390/jcm9051456. PMID 32414075
- [Background] Vizza CD, Hoeper MM, Huscher D, Pittrow D, Benjamin N, Olsson KM, Ghofrani HA, Held M, Klose H, Lange T, Rosenkranz S, Dumitrescu D, Badagliacca R, Claussen M, Halank M, Vonk-Noordegraaf A, Skowasch D, Ewert R, Gibbs JSR, Delcroix M, Skride A, Coghlan G, Ulrich S, Opitz C, Kaemmerer H, Distler O, Grunig E. Pulmonary Hypertension in Patients With COPD: Results From the Comparative, Prospective Registry of Newly Initiated Therapies for Pulmonary Hypertension (COMPERA). Chest. 2021 Aug;160(2):678-689. doi: 10.1016/j.chest.2021.02.012. Epub 2021 Feb 11. PMID 33581097
- [Background] Rosenkranz S, Pausch C, Coghlan JG, Huscher D, Pittrow D, Grunig E, Staehler G, Vizza CD, Gall H, Distler O, Delcroix M, Ghofrani HA, Ewert R, Kabitz HJ, Skowasch D, Behr J, Milger K, Halank M, Wilkens H, Seyfarth HJ, Held M, Scelsi L, Neurohr C, Vonk-Noordegraaf A, Ulrich S, Klose H, Claussen M, Eisenmann S, Schmidt KH, Remppis BA, Skride A, Jureviciene E, Gumbiene L, Miliauskas S, Loffler-Ragg J, Lange TJ, Olsson KM, Hoeper MM, Opitz C. Risk stratification and response to therapy in patients with pulmonary arterial hypertension and comorbidities: A COMPERA analysis. J Heart Lung Transplant. 2023 Jan;42(1):102-114. doi: 10.1016/j.healun.2022.10.003. Epub 2022 Oct 13. PMID 36333206
- [Background] Hoeper MM, Dwivedi K, Pausch C, Lewis RA, Olsson KM, Huscher D, Pittrow D, Grunig E, Staehler G, Vizza CD, Gall H, Distler O, Opitz C, Gibbs JSR, Delcroix M, Park DH, Ghofrani HA, Ewert R, Kaemmerer H, Kabitz HJ, Skowasch D, Behr J, Milger K, Lange TJ, Wilkens H, Seyfarth HJ, Held M, Dumitrescu D, Tsangaris I, Vonk-Noordegraaf A, Ulrich S, Klose H, Claussen M, Eisenmann S, Schmidt KH, Swift AJ, Thompson AAR, Elliot CA, Rosenkranz S, Condliffe R, Kiely DG, Halank M. Phenotyping of idiopathic pulmonary arterial hypertension: a registry analysis. Lancet Respir Med. 2022 Oct;10(10):937-948. doi: 10.1016/S2213-2600(22)00097-2. Epub 2022 Jun 28. PMID 35777416
- [Background] Hoeper MM, Pausch C, Olsson KM, Huscher D, Pittrow D, Grunig E, Staehler G, Vizza CD, Gall H, Distler O, Opitz C, Gibbs JSR, Delcroix M, Ghofrani HA, Park DH, Ewert R, Kaemmerer H, Kabitz HJ, Skowasch D, Behr J, Milger K, Halank M, Wilkens H, Seyfarth HJ, Held M, Dumitrescu D, Tsangaris I, Vonk-Noordegraaf A, Ulrich S, Klose H, Claussen M, Lange TJ, Rosenkranz S. COMPERA 2.0: a refined four-stratum risk assessment model for pulmonary arterial hypertension. Eur Respir J. 2022 Jul 7;60(1):2102311. doi: 10.1183/13993003.02311-2021. Print 2022 Jul. PMID 34737226
- [Background] Distler O, Ofner C, Huscher D, Jordan S, Ulrich S, Stahler G, Grunig E, Held M, Ghofrani HA, Claussen M, Lange TJ, Klose H, Rosenkranz S, Vonk-Noordegraaf A, Vizza CD, Delcroix M, Opitz C, Pausch C, Scelsi L, Neurohr C, Olsson KM, Coghlan JG, Halank M, Skowasch D, Behr J, Milger K, Remppis BA, Skride A, Jureviciene E, Gumbiene L, Miliauskas S, Loffler-Ragg J, Wilkens H, Pittrow D, Hoeper MM, Ewert R. Treatment strategies and survival of patients with connective tissue disease and pulmonary arterial hypertension: a COMPERA analysis. Rheumatology (Oxford). 2024 Apr 2;63(4):1139-1146. doi: 10.1093/rheumatology/kead360. PMID 37462520
- [Background] Schmidt KH, Milger K, Pausch C, Huscher D, Pittrow D, Grunig E, Staehler G, Gall H, Distler O, Skowasch D, Halank M, Wilkens H, Held M, Klose H, Hoeper MM. Trends in COVID-19-associated mortality in patients with pulmonary hypertension: a COMPERA analysis. Eur Respir J. 2023 Apr 27;61(4):2202440. doi: 10.1183/13993003.02440-2022. Print 2023 Apr. PMID 37105586
- [Derived] Kaemmerer AS, Gorenflo M, Huscher D, Pittrow D, Ewert P, Pausch C, Delcroix M, Ghofrani HA, Hoeper MM, Kozlik-Feldmann R, Skride A, Stahler G, Vizza CD, Jureviciene E, Jancauskaite D, Gumbiene L, Ewert R, Dahnert I, Held M, Halank M, Skowasch D, Klose H, Wilkens H, Milger K, Jux C, Koestenberger M, Scelsi L, Brunnemer E, Hofbeck M, Ulrich S, Vonk Noordegraaf A, Lange TJ, Bruch L, Konstantinides S, Claussen M, Loffler-Ragg J, Wirtz H, Apitz C, Neidenbach R, Freilinger S, Nemes A, Opitz C, Grunig E, Rosenkranz S. Medical treatment of pulmonary hypertension in adults with congenital heart disease: updated and extended results from the International COMPERA-CHD Registry. Cardiovasc Diagn Ther. 2021 Dec;11(6):1255-1268. doi: 10.21037/cdt-21-351. PMID 35070795
- [Derived] Hoeper MM, Behr J, Held M, Grunig E, Vizza CD, Vonk-Noordegraaf A, Lange TJ, Claussen M, Grohe C, Klose H, Olsson KM, Zelniker T, Neurohr C, Distler O, Wirtz H, Opitz C, Huscher D, Pittrow D, Gibbs JS. Pulmonary Hypertension in Patients with Chronic Fibrosing Idiopathic Interstitial Pneumonias. PLoS One. 2015 Dec 2;10(12):e0141911. doi: 10.1371/journal.pone.0141911. eCollection 2015. PMID 26630396
- [Derived] Kaemmerer H, Gorenflo M, Hoeper M, Huscher D, Ewert P, Pittrow D. [Pulmonary arterial hypertension in patients with congenital heart disease: current issues and health care situation]. Dtsch Med Wochenschr. 2013 Jun;138(23):1247-52. doi: 10.1055/s-0033-1343189. Epub 2013 May 29. German. PMID 23720182
- See also: COMPERA website — https://www.compera.org/